CLINICAL TRIAL: NCT05845411
Title: Impact of a Nutritional Intervention Based on Mindful Eating on the Eating Behavior of Individuals Living With Overweight and Obesity
Brief Title: Mindful Eating for Eating Behavior Individuals Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Maria Fernanda Souza Moreira, RD, MSc, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE46133421100005345
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Overweight and Obesity; Behavior, Eating; Feeding Patterns
Keywords: Mindfulness; Mindful Eating; Weight management;
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A group of 30 people will participate in 8 fortnightly virtual group sessions for 4 months, where the subject of Mindful Eating will be addressed. Participants will be encouraged to share their eating experiences, reflect and discuss the above, and engage in formal and non-formal mindfulness eating practices (meditation, eating slowly, observing thoughts, and being present at meal times) between sessions.
  Interventions: Behavioral: Mindful Eating
- Control (Active Comparator): A group of 30 people will have 8 fortnightly, virtual, and individual consultations for 4 months. They will receive a hypocaloric diet (reduction of approximately 500kcal per day in total energy expenditure) and food and nutrition education. The food plan will be monitored in each meeting, and a theme of food and nutrition education will be worked on, based on the Food Guide for the Brazilian Population, through expository content. A virtual folder of all subjects taught will be provided.
  Interventions: Other: Standard dietary treatment

INTERVENTIONS:
Behavioral: Mindful Eating — Nutritional advice through expository content, group discussion, and exchange of experiences on self-knowledge, food awareness, and relationship with food and the body.
  Arms: Intervention
Other: Standard dietary treatment — Hypocaloric dietary prescription and nutritional education.
  Arms: Control

SUMMARY:
This clinical trial aims to compare the effect of a nutritional intervention based on Mindful Eating, with standard dietary treatment, in changing the eating behavior of overweight individuals.

DETAILED DESCRIPTION:
This clinical trial aims to compare the effect of a nutritional intervention based on Mindful Eating, with standard dietary treatment, in changing the eating behavior of overweight individuals. The main questions to answer are:

* What is the effect of the intervention on the domains of eating behavior (emotional eating, cognitive restriction, and lack of food control - assessed by the Three-Factor Eating Questionnaire R21)? ,
* Assess the effect of the intervention on weight and BMI.
* Evaluate the relationship between eating behavior domains before and after the intervention.

Participants in the intervention group will participate in eight sessions of a virtual therapeutic group, with up to fifteen individuals, every fifteen days, in which the theme of Mindful Eating and eating behavior will be worked. Participants will be encouraged to undertake the following:

* self-knowledge exercises between one session and another.
* mindfulness meditations daily. No dietary plan will be provided.

The researchers will compare the results with a control group, which will receive eight individual, fortnightly, and virtual consultations of conventional dietary treatment, which will provide:

* dietary plan for weight reduction, according to current guidelines.
* six food and nutrition education sessions based on the Food Guide for the Brazilian Population.

ELIGIBILITY:
Inclusion Criteria:

* body mass index greater than or equal to 25 kg/m²,
* internet access,
* availability to participate in 8 virtual meetings.

Exclusion Criteria:

* volunteers using pharmacotherapy for obesity,
* pregnancy,
* lactation,
* cognitive conditions, self-reported neurological or psychiatric disorders that prevent participation in the study,
* decompensated thyroid disorders, and
* who have undergone bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in eating behavior | Four months
  Sub-divided into domains: uncontrolled eating (UE), cognitive restriction (CR), and emotional eating (EE).

SECONDARY OUTCOMES:
Body weight | Four months
  in kilos
Body Mass Index - BMI | Four months
  in kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernanda Souza Moreira, MSc, Principal Investigator — Federal University of Health Sciences of Porto Alegre; Fernanda Michielin Busnello, PhD, Study Director — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Moreira MFS, de Azevedo BEF, Beretta MV, Busnello FM. Nutritional Counseling Based on Mindful Eating for the Eating Behavior of People Living with Overweight and Obesity: A Randomized Clinical Trial. Nutrients. 2024 Dec 20;16(24):4388. doi: 10.3390/nu16244388. PMID 39771009